CLINICAL TRIAL: NCT02503111
Title: A Randomized Controlled, Open-label Trial Examining the Efficacy, Safety, and Tolerability of Ablative Therapies for High-grade Anal Dysplasia Versus Observation Alone in HIV-positive Men Who Have Sex With Men (MSM)
Brief Title: The HPV-SAVE Study Team: HPV Screening and Vaccine Evaluation in Men Who Have Sex With Men
Acronym: HPV-SAVE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Results from ANCHOR study showed benefit of Treatment over Surveillance in preventing anal cancer.
  That study was similar to the current one.
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Ontario HIV Treatment Network (Network); CIHR Canadian HIV Trials Network (Network); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Irving Salit, Immunodeficiency Clinic Director, Toronto General Hospital, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTN 292B
Record Dates: First submitted 2015-07-10; First posted 2015-07-20 (Estimated); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Anal Dysplasia; Human Papillomavirus; Anal Cancer
Keywords: Men who have sex with men; Human immunodeficiency virus; Human papillomavirus; Anal intraepithelial neoplasia; Squamous cell carcinoma; High-resolution anoscopy; Anal cancer; High-risk oncogenic; Intraepithelial lesion; Low-risk non-oncogenic; Dysplasia; High-grade squamous intraepithelial lesion; Low-grade squamous intraepithelial lesion; Ablative therapy; Electrocautery; Infrared coagulation; Active surveillance
MeSH Terms: conditions — Anus Neoplasms; Homosexuality; Acquired Immunodeficiency Syndrome; Carcinoma, Squamous Cell; Squamous Intraepithelial Lesions | interventions — Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ablative therapy (Experimental): Ablative therapy involving electrocautery (EC) will occur for participants with AIN-2 and AIN-3. The Hyfrecator ® 2000 Electrosurgical System will be used for EC therapy.
  Interventions: Device: The Hyfrecator ® 2000 Electrosurgical System
- Active Surveillance (Active Comparator): The control arm includes active surveillance with observation alone; no treatment in AIN-2 and -3.
  Interventions: Other: Observation Alone

INTERVENTIONS:
Device: The Hyfrecator ® 2000 Electrosurgical System — Lesion is ablated by the The Hyfrecator ® 2000 Electrosurgical System. During electrocautery (EC) with The Hyfrecator, a gentle brushing technique occurs and the tissue is removed with forceps.
  Other Names: EC
  Arms: Ablative therapy
Other: Observation Alone — No treatment to AIN-2 or AIN-3, only active surveillance.
  Arms: Active Surveillance

SUMMARY:
Human papillomavirus (HPV) is the most common sexually transmitted infection worldwide. Infection by certain high-risk oncogenic types of HPV (HR-HPV) is the major cause of several cancers in men, notably squamous cell carcinoma (SCC) of the anal canal. Rates of anal infection with these HR-HPV strains and the resultant high-grade anal dysplasia and anal cancer are much higher in men who have sex with men (MSM) than in the general population. Co-infection with human immunodeficiency virus (HIV) further amplifies this burden, making the rates of anal SCC in HIV-positive MSM higher than the historic rates of cervical cancer prior to the adoption of routine cervical cytology screening. Despite these alarming statistics, there are no established protocols for optimal screening and treatment of anal HPV and cancer precursors, nor has there been any widespread rollout of organized screening programs anywhere in Canada. Further, not only does HPV directly cause significant disease in these men, but there is growing epidemiologic evidence that HPV infection may enhance sexual transmission of HIV. These significant knowledge gaps translate into fundamental deficiencies in care for HIV-positive MSM.

The HPV Screening and Vaccine Evaluation in MSM (HPV-SAVE) study team will recruit a large group of MSM from various Ontario and Vancouver clinics, in order to carry out a number of different studies. The HPV-SAVE team brings together community and internationally-recognized experts in HPV and HIV disease and mucosal immunology, to better define the optimal approaches for primary and secondary prevention and treatment of HPV-associated anal disease among HIV-positive MSM, and to explore biological mechanistic evidence regarding the potential role of HPV as a co-factor for HIV transmission. This will yield critical information which can lead to improvement in the health of MSM, and will provide a foundation on which to build further, large-scale screening and treatment trials on a national level. The primary aim of the current study is to systematically compare ablative therapy versus intensive observation alone (also known as 'watchful waiting') in outcomes relating to high-grade anal dysplasia.

DETAILED DESCRIPTION:
Since the 1990s, combination antiretroviral therapy (cART) has markedly reduced HIV-related opportunistic infections and mortality [1], and increased the life expectancy of people living with HIV [2]. While acquired immune deficiency syndrome (AIDS)-defining malignancies have declined [3,4], non-AIDS defining malignancies continue to occur at higher rates in HIV-infected persons than in the general population [4]. Amongst these are cancers associated with HPV which is responsible for the vast majority of cervical cancers (itself a well-established AIDS-defining illness), and an estimated 90% of SCC of the anal canal [5]. cART not only fails to protect against anal pre-cancers and cancers [4,6,7], but the incidence of anal SCC is increasing in the cART era [6,8]. Because of this increasing burden of disease, there is an urgent need to find effective ways of preventing anal SCC in those living with HIV. This includes screening for anal cancer precursors and ablative treatment of these lesions.

Though it is infrequent at a rate of 1 per 100 000, anal SCC is on the rise in the general population [9]. It occurs at significantly higher rates in HIV-positive men - particularly among men who have sex with men (MSM) - with an estimated rate of 60 to 160 per 100 000 [4], and no evidence of slowing in the era of increased cART use [10] (See Figure 1). In fact, rates of anal cancer among HIV-infected MSM are comparable to rates of cervical cancer in women prior to the adoption of routine screening for cervical dysplasia [11]. According to data from the Public Health Agency of Canada, rates of cervical cancer in 1972 were 18 per 100 000, dropping to just under 8 per 100 000 in 2004 [12]. In addition to its etiologic association with HPV, anal cancer shares many similarities with cervical cancer. Both are squamous cell cancers occurring at the squamocolumnar junction [13,14] and both likely arise from histologically-similar dysplastic precursor lesions [15,16]. It is postulated that a critical step in anal cancer carcinogenesis is the establishment of persistent infection with oncogenic HPV in the anal canal [16]. Though the majority of HPV infections are considered transient and will eventually clear even in HIV-positive individuals [17], HIV-positive individuals have higher rates of persistent infection, especially with oncogenic HPV types [18].

Of the greater than 170 HPV types, over 50 favour the anogenital area and, on the basis of epidemiologic and phylogenetic data, these have been classified by the International Agency for Research on Cancer [19]. The vast majority of anal cancers (as well as cervical cancers) are caused by two high-risk HPV types: HPV type 16 and HPV type 18 which are responsible for 66% and 5% of anal cancers, respectively [20]. HPV lesions caused by low-risk HPV (LR-HPV) types include condylomata (commonly known as 'genital warts'), of which 90% are caused by HPV types 6 and 11 [21]. Prevention strategies for anal cancers have emerged that are analogous to strategies used in cervical cancer screening, in that the aim is to identify precursor lesions which can then be removed before progression to cancer. Screening and detection rely on a combination of anal cytology (Papanicolaou, or Pap smear), anal HPV detection and high-resolution anoscopy (HRA) which is analogous to colposcopy). Visually-directed anal biopsy during HRA is considered the gold standard for detecting dysplastic lesions such as high-grade anal intraepithelial neoplasia (HGAIN; typically graded as AIN-2 or -3) [16,22]. Anal cytology is generally used as a screening test to determine whether HRA is needed; however, cytology is an imperfect predictor of intra-anal HGAIN. Despite the clear evidence indicating the benefit of screening and treatment procedures in cervical cancer screening, no large rigorous studies have been performed to assess such strategies in anal cancer prevention in men or women.

ELIGIBILITY:
Inclusion Criteria:

* Males, aged ≥18 years at baseline;
* Identify as a man who has sex with a men (MSM);
* HIV-positive; laboratory documentation of HIV-1 infection;
* For those on combination antiretroviral therapy (cART), the participant must be on a stable regimen;
* An ability to give informed consent;
* An ability to attend clinic for follow-up, including possible HRA and biopsy;
* AIN-2 or -3 found on biopsy of anal canal lesion(s);
* Willingness to be randomized to undergo ablative therapy or active surveillance.

Exclusion Criteria:

* Current or prior history of cancer of the anogenital regions (e.g. penile, anal, or rectal).;
* Previous treatment of high grade dysplasia;

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2015-11; Primary Completion 2021-11-01 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Anal dysplasia treatment on a per-patient basis | Participants will be followed after post-treatment completion, an expected average of 6 months
  Histologic resolution of high-grade AIN after treatment completion, with ablative therapies or surveillance alone. Resolution of high-grade AIN will be defined as histologic diagnosis of AIN-1 or normal at the post treatment HRA.

SECONDARY OUTCOMES:
Resolution of high-grade AIN at 3 and 6 months after randomization, on a per-lesion basis | Participants will be followed after post-treatment completion, an expected average of 6 months
  Resolution of high-grade AIN after treatment on a per-lesion basis. Histologic resolution of high-grade AIN after treatment completion, with ablative therapies or surveillance alone. Resolution of high-grade AIN will be defined as histologic diagnosis of AIN-1 or normal at the post treatment HRA.
Recurrence rates of high-grade AIN | Participants will be followed post-treatment completion, at 12, 24 and 36 months after randomization
  Recurrence rates of high-grade AIN following ablative therapy on a per lesion basis.
Number of participants with adverse events | Participants will be followed after post-treatment completion, an expected average of 36 months
  Number of participants assessed on safety, tolerability and acceptability of the different intervention arms and the different treatments in the ablative therapies arms. Evaluation of adverse events and questionnaire-assessed acceptability by intervention arms and ablative treatment type.
Acceptability of treatment | Within 6 months of randomization
  Questionnaire-assessed acceptability by intervention arm

CONTACTS AND LOCATIONS:
Overall Officials: Irving Salit, MD, Principal Investigator — Toronto General Hospital, University Health Network
Locations (4):
- Canada (4):
  - BC Centre for Disease Control, Vancouver, British Columbia
  - University of British Columbia, Vancouver, British Columbia
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario

REFERENCES:
- [Background] Palella FJ Jr, Delaney KM, Moorman AC, Loveless MO, Fuhrer J, Satten GA, Aschman DJ, Holmberg SD. Declining morbidity and mortality among patients with advanced human immunodeficiency virus infection. HIV Outpatient Study Investigators. N Engl J Med. 1998 Mar 26;338(13):853-60. doi: 10.1056/NEJM199803263381301. PMID 9516219
- [Background] Lohse N, Hansen AB, Pedersen G, Kronborg G, Gerstoft J, Sorensen HT, Vaeth M, Obel N. Survival of persons with and without HIV infection in Denmark, 1995-2005. Ann Intern Med. 2007 Jan 16;146(2):87-95. doi: 10.7326/0003-4819-146-2-200701160-00003. PMID 17227932
- [Background] Patel P, Hanson DL, Sullivan PS, Novak RM, Moorman AC, Tong TC, Holmberg SD, Brooks JT; Adult and Adolescent Spectrum of Disease Project and HIV Outpatient Study Investigators. Incidence of types of cancer among HIV-infected persons compared with the general population in the United States, 1992-2003. Ann Intern Med. 2008 May 20;148(10):728-36. doi: 10.7326/0003-4819-148-10-200805200-00005. PMID 18490686
- [Background] Silverberg MJ, Chao C, Leyden WA, Xu L, Tang B, Horberg MA, Klein D, Quesenberry CP Jr, Towner WJ, Abrams DI. HIV infection and the risk of cancers with and without a known infectious cause. AIDS. 2009 Nov 13;23(17):2337-45. doi: 10.1097/QAD.0b013e3283319184. PMID 19741479
- [Background] Parkin DM, Bray F. Chapter 2: The burden of HPV-related cancers. Vaccine. 2006 Aug 31;24 Suppl 3:S3/11-25. doi: 10.1016/j.vaccine.2006.05.111. PMID 16949997
- [Background] Crum-Cianflone NF, Hullsiek KH, Marconi VC, Ganesan A, Weintrob A, Barthel RV, Agan BK; Infectious Disease Clinical Research Program HIV Working Group. Anal cancers among HIV-infected persons: HAART is not slowing rising incidence. AIDS. 2010 Feb 20;24(4):535-43. doi: 10.1097/QAD.0b013e328331f6e2. PMID 19926961
- [Background] van Leeuwen MT, Vajdic CM, Middleton MG, McDonald AM, Law M, Kaldor JM, Grulich AE. Continuing declines in some but not all HIV-associated cancers in Australia after widespread use of antiretroviral therapy. AIDS. 2009 Oct 23;23(16):2183-90. doi: 10.1097/QAD.0b013e328331d384. PMID 19734774
- [Background] Piketty C, Selinger-Leneman H, Grabar S, Duvivier C, Bonmarchand M, Abramowitz L, Costagliola D, Mary-Krause M; FHDH-ANRS CO 4. Marked increase in the incidence of invasive anal cancer among HIV-infected patients despite treatment with combination antiretroviral therapy. AIDS. 2008 Jun 19;22(10):1203-11. doi: 10.1097/QAD.0b013e3283023f78. PMID 18525266
- [Background] Chiao EY, Krown SE, Stier EA, Schrag D. A population-based analysis of temporal trends in the incidence of squamous anal canal cancer in relation to the HIV epidemic. J Acquir Immune Defic Syndr. 2005 Dec 1;40(4):451-5. doi: 10.1097/01.qai.0000159669.80207.12. PMID 16280701
- [Background] Piketty C, Selinger-Leneman H, Bouvier AM, Belot A, Mary-Krause M, Duvivier C, Bonmarchand M, Abramowitz L, Costagliola D, Grabar S. Incidence of HIV-related anal cancer remains increased despite long-term combined antiretroviral treatment: results from the french hospital database on HIV. J Clin Oncol. 2012 Dec 10;30(35):4360-6. doi: 10.1200/JCO.2012.44.5486. Epub 2012 Oct 22. PMID 23091098
- [Background] Qualters JR, Lee NC, Smith RA, Aubert RE. Breast and cervical cancer surveillance, United States, 1973-1987. MMWR CDC Surveill Summ. 1992 Apr 24;41(2):1-7. PMID 1594012
- [Background] Public Health Agency of Canada. Available at: http://www.phac-aspc.gc.ca/cd- mc/cancer/cervical_cancer_figures-cancer_du_col_uterus-eng.php. Accessed on: 28 July 2014.
- [Background] de Ruiter A, Mindel A. Anal intraepithelial neoplasia. Eur J Cancer. 1991;27(11):1343-5. doi: 10.1016/0277-5379(91)90004-w. No abstract available. PMID 1660290
- [Background] Bjorge T, Engeland A, Luostarinen T, Mork J, Gislefoss RE, Jellum E, Koskela P, Lehtinen M, Pukkala E, Thoresen SO, Dillner J. Human papillomavirus infection as a risk factor for anal and perianal skin cancer in a prospective study. Br J Cancer. 2002 Jul 1;87(1):61-4. doi: 10.1038/sj.bjc.6600350. PMID 12085257
- [Background] Watson AJ, Smith BB, Whitehead MR, Sykes PH, Frizelle FA. Malignant progression of anal intra-epithelial neoplasia. ANZ J Surg. 2006 Aug;76(8):715-7. doi: 10.1111/j.1445-2197.2006.03837.x. PMID 16916390
- [Background] Palefsky JM, Holly EA, Hogeboom CJ, Ralston ML, DaCosta MM, Botts R, Berry JM, Jay N, Darragh TM. Virologic, immunologic, and clinical parameters in the incidence and progression of anal squamous intraepithelial lesions in HIV-positive and HIV-negative homosexual men. J Acquir Immune Defic Syndr Hum Retrovirol. 1998 Apr 1;17(4):314-9. doi: 10.1097/00042560-199804010-00004. PMID 9525431
- [Background] Giuliano AR, Lu B, Nielson CM, Flores R, Papenfuss MR, Lee JH, Abrahamsen M, Harris RB. Age-specific prevalence, incidence, and duration of human papillomavirus infections in a cohort of 290 US men. J Infect Dis. 2008 Sep 15;198(6):827-35. doi: 10.1086/591095. PMID 18657037
- [Background] Trottier H, Franco EL. The epidemiology of genital human papillomavirus infection. Vaccine. 2006 Mar 30;24 Suppl 1:S1-15. doi: 10.1016/j.vaccine.2005.09.054. PMID 16406226
- [Background] Bouvard V, Baan R, Straif K, Grosse Y, Secretan B, El Ghissassi F, Benbrahim-Tallaa L, Guha N, Freeman C, Galichet L, Cogliano V; WHO International Agency for Research on Cancer Monograph Working Group. A review of human carcinogens--Part B: biological agents. Lancet Oncol. 2009 Apr;10(4):321-2. doi: 10.1016/s1470-2045(09)70096-8. No abstract available. PMID 19350698
- [Background] Hoots BE, Palefsky JM, Pimenta JM, Smith JS. Human papillomavirus type distribution in anal cancer and anal intraepithelial lesions. Int J Cancer. 2009 May 15;124(10):2375-83. doi: 10.1002/ijc.24215. PMID 19189402
- [Background] Kjaer SK, Tran TN, Sparen P, Tryggvadottir L, Munk C, Dasbach E, Liaw KL, Nygard J, Nygard M. The burden of genital warts: a study of nearly 70,000 women from the general female population in the 4 Nordic countries. J Infect Dis. 2007 Nov 15;196(10):1447-54. doi: 10.1086/522863. Epub 2007 Oct 31. PMID 18008222
- [Background] Jay N, Berry JM, Hogeboom CJ, Holly EA, Darragh TM, Palefsky JM. Colposcopic appearance of anal squamous intraepithelial lesions: relationship to histopathology. Dis Colon Rectum. 1997 Aug;40(8):919-28. doi: 10.1007/BF02051199. PMID 9269808